CLINICAL TRIAL: NCT02563210
Title: Interrupter Technique and Plethysmography Airway Resistance Measurement: Comparison of These Two Techniques for the Diagnosis of Airway Obstruction Diagnosis and Bronchodilation Response in Children 3 to 6 Years of Age
Brief Title: Airway Resistance Measurement in Children 3 to 6 Years of Age
Acronym: ARC36
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARC 36 (RB 15.181)
Record Dates: First submitted 2015-09-15; First posted 2015-09-30 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2017-06

CONDITIONS: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- airway resistance measurement (Experimental): interruption and plethysmography techniques airway resistance measurement at each routine visit
  Interventions: Other: airway resistance measurement

INTERVENTIONS:
Other: airway resistance measurement — assessment of airway resistance

SUMMARY:
In preschool aged children, the most suitable techniques to assess airway obstruction is debit interruption technic (Rint) and plethysmographic measure of specific airway resistance (sRaw). Even if Rint is easily and routinely performed, it also includes a component of lung tissue and chest wall resistance as well as respiratory tissue viscoelasticity. sRaw seems to be better for discriminating airway obstruction. These two techniques will be compared in terms of concordance in the diagnosis of pulmonary obstruction and bronchodilator response.

ELIGIBILITY:
Inclusion Criteria:

* Child 3 to 6 years aged

Exclusion Criteria:

* Height below 90 centimeters
* Opposition to participation

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-05-29 (Actual)

PRIMARY OUTCOMES:
airway resistance measure by interruption technique (Rint) | Day one
  Rint is performed using Spiroteq Dyn'R during a 100 ms occlusion and calculated using the linear back extrapolation method

SECONDARY OUTCOMES:
measure of bronchodilator response | Day one
  Bronchodilator response is assessed with Rint and sRaw measurement

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Agnès METGES, Pr, Principal Investigator — University Hospital of Brest
Locations (1):
- CHRU de Brest, Brest, France

REFERENCES:
- [Derived] Mauger-Hamel P, Du Boisbaudry C, Leon K, Alavi Z, Giroux-Metges MA. Relationship between baseline and post-bronchodilator interrupter resistance and specific airway resistance in preschool children. Ann Allergy Asthma Immunol. 2020 Apr;124(4):366-372. doi: 10.1016/j.anai.2020.01.003. Epub 2020 Jan 13. PMID 31945475